CLINICAL TRIAL: NCT01979432
Title: The Cognitive and Cardiovascular Health in the Elderly Study
Acronym: COACHES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: I11014
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Diseases
Keywords: Alzheimer, cognitive diseases, Ankle-to-brachial index
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cardiovascular evaluation (Other): Measure of the index of systolic pressure Echo doppler Echography Measure of the speed of the wave of pulse and the central pressure
  Interventions: Other: Cardiovascular evaluation

INTERVENTIONS:
Other: Cardiovascular evaluation

SUMMARY:
The main objective of this study is to look for the interest forecast of the IPS as infra-clinical cardiovascular marker in the prediction of a change of the cognitive functions (MCI) at the elderly of 70 and more years old without clinical cardiovascular pathology.

ELIGIBILITY:
Inclusion Criteria:

* free-living community-dwelling men and women aged ≥ 70 years,
* subjects free of clinical CVD related to atherosclerosis
* preserved basic activities of daily living (ADL = 6)
* without cognitive impairment (MMSE≥24)

Exclusion Criteria:

* subjects with clinical history of any of the following CVD diseases : coronary artery disease (angina, myocardial infarction, coronary revascularization), cerebrovascular disease (stroke, TIA, carotid revascularization), clinical peripheral artery disease (claudication, critical limb ischemia)
* subjects with neurodegenerative, locomotor and ophtalmological diseases unable to perform the cognitive tests
* subjects unable to give written informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12-12 (Actual); Study Completion 2015-12-12 (Actual)

PRIMARY OUTCOMES:
Incident "MCI" according to the following criteria | one time point
  (1) cognitive complaint (self-reported and/or informant) ; (2) preserved basic activities of daily living (ADL) ; (3) cognitive impairment (not normal for age and education) or decline in cognition evidenced by performance on objective cognitive tasks defined as a test performance <1.0 standard deviations below the mean of the reference group ; (4) preserved general cognitive functioning and (5) absence of dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Limoges, Limoges, France